CLINICAL TRIAL: NCT05568966
Title: Collection of Venous and Capillary Blood Samples for the Research, Optimisation and Calibration of New Diagnostic Devices 2
Brief Title: Collection of Blood Samples for New Diagnostic Devices 2
Acronym: NOVEL-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LumiraDx UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S-CLIN-PROT-00025
Record Dates: First submitted 2022-09-21; First posted 2022-10-06 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Embolism and Thrombosis; Cardiovascular; Renal; Inflammation; Infections
MeSH Terms: conditions — Embolism and Thrombosis; Inflammation; Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood Draw (Experimental): Venous blood draw up to 24mL and/or 6 capillary fingersticks
  Interventions:
  Diagnostic Test: Venepuncture Diagnostic Test: Fingerstick
  Interventions: Diagnostic Test: Venous blood draw; Diagnostic Test: Fingerstick

INTERVENTIONS:
Diagnostic Test: Venous blood draw — Venepuncture to draw up to 24mL of venous blood.
Diagnostic Test: Fingerstick — Capillary blood draw

SUMMARY:
To research and develop new state of the art diagnostic biomarkers on the LumiraDx Platform that are comparable to the approved gold standard reference methods and will radically enhance clinicians and patients ability to monitor health conditions and improve outcomes by delivering the results near patient at the point of care.

DETAILED DESCRIPTION:
This is a comparative research study to research, optimise and develop new state of the art diagnostic biomarkers on the LumiraDx Platform that will radically enhance clinicians and patients ability to monitor chronic health conditions which improve outcomes at the point of care and that are comparable to gold standard reference methods. The LumiraDx POC Platform consists of an in vitro diagnostic instrument, used with single use test strips for different disease biomarkers. This next generation point of care device is intended to allow multiple tests to be performed on the same platform for blood, plasma, serum, swab, and urine samples.

Research activities will be completed on blood samples collected from a maximum of 20,000 patients to assess the performance of the new biomarkers undergoing research. Patients will include those presenting at a medical unit (including but not limited to A&E departments, hospital wards, or out-patient clinics) to their care team, in order to obtain a range of values for research of the new biomarkers on the LumiraDx system. Participants will include those who are expected to have (but are not limited to) biomarkers for diseases areas including embolism, infection or inflammation, cardiovascular, and renal cohorts.

Each patient must give appropriate written informed consent and satisfy all the inclusion/exclusion criteria prior to any study procedures. Patient participation in this study will take a maximum of 45 minutes of the patient's time. Patients presenting for a subsequent clinic visit or admission may be approached to participate in the study again, a maximum of 24mL of venous whole blood and up to 6 capillary fingersticks (obtained with a high flow lancet) may be collected from each patient within a three month period. Where possible, study samples should be taken at the same time as any standard of care blood draws or from patients with a cannula in-situ, a separate study venipuncture is not a requirement for this protocol. Study samples will be used for research, evaluation, optimisation and development activities into new biomarkers on the LumiraDx Platform in comparison with the gold standard reference method for the disease area to ensure comparable performance. Samples may also be used for troubleshooting and calibrating LumiraDx assays developed.

Sample collection will be separated into 2 phases depending upon the research needs. Patients can participate in both phases:

Phase 1: Only venous blood samples will be drawn by the HCP. These samples will be tested on the LumiraDx System and/or device(s) under development and also tested on the appropriate reference method for comparison. This testing may occur at the clinical site and/or at LumiraDx UK Ltd.

Phase 2: Venous blood samples and capillary fingerstick samples will be collected by the HCP. These samples may be tested on the LumiraDx Platform and also tested on the appropriate reference method for comparison. The fingerstick samples will be tested on the LumiraDx device. The processing of samples may occur at the clinical site and/or at LumiraDX UK Ltd.

The samples will be identified by patient identification number, anonymising the patient's identifiable information. These blood samples will be sent to LumiraDx UK Ltd for storage and future testing. No genetic testing will be carried out on samples. Samples may also be used to research, optimise, develop, modify and calibrate products and platforms for measuring biomarkers including, but not limited to, Troponin, NT-pro BNP, BNP, CK-MB, D-Dimer, NGAL, Cystatin C, Myoglobin, Galectin-3, CRP, AST, ALT, Lipids, Coagulation, Prolactin, and Beta-hCG.

Patients who reattend or are admitted to the medical unit (including but not limited to A&E departments, hospital wards or out-patient clinics) may be asked for further sampling. A total of 24mL and 6 capillary fingersticks (obtained using high flow lancets) will not be exceeded over the three month period from consent, patients may opt out of further contact. Any patient reattending three months post consent will be treated as a new patient.

Data will be recorded on the Case Report Forms. The patient demographics data collected may include: age; sex; ethnicity, pregnancy status, NYHA classification, current medications at time of blood collection including their indications, significant medical history, relevant local blood test results, reason(s) for presenting, and confirmed diagnosis.

ELIGIBILITY:
Inclusion Criteria

* Subject 18 years of age.
* Willing and able to provide written informed consent and comply with study procedures.
* Patients attending a definitive care team with research capabilities which has been enroled in this collection study.
* Patients who can read and understand written English.
* The subject must present as one of the following cohorts:

  1. Group A - Embolism Cohort - Patients presenting with symptoms indicative of thromboembolic events.
  2. Group B - Infection or Inflammation Cohort - Patients presenting with symptoms indicative of infection or inflammatory disorders.
  3. Group C - Cardiovascular Cohort - Patients presenting with symptoms indicative of heart failure or acute coronary syndrome.
  4. Group D - Renal Cohort - Patients presenting with symptoms indicative of renal disorders.
  5. Group E - Other Cohort. - Patients who are not eligible for any of the above groups.

Exclusion Criteria

* Subject <18 years of age.
* Vulnerable populations deemed inappropriate for the study by the sites Principal Investigator.
* Patients who have previously been enroled in any LumiraDx NOVEL study in the past 3 months and re-entry would breach the 24mL and or 6 fingersitck maximums.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Measurement of blood samples from patients with infection, cardiovascular disease, embolism or renal disease in a reference method and in a novel LumiraDx method. | Up to 5 years
  Measurement of blood samples in a reference method and in a novel LumiraDx method to assess accuracy of the LumiraDx method in patients with infection, cardiovascular disease, embolism or renal disease. Accuracy will be assessed by regression analysis against a reference method.
Multiple measurements of blood samples from patients with infection, cardiovascular disease, embolism or renal disease in a novel LumiraDx method. | Up to 5 years
  Multiple measurements of blood samples in a novel LumiraDx method to assess precision of the method in patients with infection, cardiovascular disease, embolism or renal disease. Precision will be assessed by coefficient of variation (%CV) estimates.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Gardner, Principal Investigator — NHS National Waiting Times Centre Board; Alasdair Gray, Principal Investigator — NHS Lothian; Allan Cameron, Principal Investigator — NHS Greater Glasgow & Clyde; David Lowe, Principal Investigator — NHS Greater Glasgow & Clyde; Santosh Bongale, Principal Investigator — NHS Greater Glasgow & Clyde; Fiona Hunter, Principal Investigator — NHS Lanarkshire
Locations (7):
- United Kingdom (7):
  - University Hospital Monklands, Airdrie, Scotland
  - Royal Infirmary of Edinburgh, Edinburgh, Scotland
  - St John's Hospital, Edinburgh, Scotland
  - Glasgow Royal Infirmary, Glasgow, Scotland
  - Queen Elizabeth University Hospital, Glasgow, Scotland
  - Golden Jubilee National Hospital, Glasgow, Scotland
  - Royal Alexandra Hospital, Paisley, Scotland

IPD SHARING:
Plan to Share IPD: No